CLINICAL TRIAL: NCT07136454
Title: Expanded Access/Compassionate Use of Rugonersen in Patients With Angelman Syndrome
Status: Available | Type: Expanded Access
Sponsor: Oak Hill Bio Ltd (Industry)
Collaborators: Early Access Care LLC (Unknown)
Responsible Party: Sponsor
Other Study IDs: OHB-EAP
Record Dates: First submitted 2025-08-14; First posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Angelman Syndrome
MeSH Terms: conditions — Angelman Syndrome

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: Rugonersen — Rugonersen is a selective synthetic 20-mer antisense oligonucleotide (ASO).

SUMMARY:
For a patient to be considered for this EAP, they must have consented to participate in the TANGELO Optional Open-label Extension (OOE), and continue to meet the inclusion/ exclusion criteria and have not received any other investigational drug for the treatment of AS between the last dose of the TANGELO OOE and the first dose in the EAP.

The Physician making the request for expanded access considers continued treatment via the EAP with rugonersen to be a suitable treatment option for the patient under consideration.

DETAILED DESCRIPTION:
The goal of this EAP is to make rugonersen available to patients who have previously consented to participate in the TANGELO Optional Open-Label Extension (OOE).

Eligibility reassessment is required for patients who are entering the EAP after they have completed a final visit in the TANGELO study. The purpose of the reassessment is to ensure that the patient continues to meet the eligibility criteria. The relevant assessments to confirm eligibility (i.e., coagulation, platelets, renal function) are part of pre-dosing assessment and can be conducted prior to EAP dosing either on the day before dosing or on the dosing day.

An updated medical history for participants should be completed prior to entering the EAP.

For the EAP the dose regimen will be 120 mg administered every 16 weeks.

ELIGIBILITY:
For a patient to be considered for this EAP, they must have consented to participate in the TANGELO Optional Open-label Extension (OOE) and, haven't deviated from any of the inclusion/ exclusion criteria and have not received any other investigational drug for the treatment of AS between the last dose of the TANGELO OOE and the first dose in the EAP.

The Physician making the request for expanded access considers continued treatment via the EAP with rugonersen to be a suitable treatment option for the patient under consideration.

Inclusion Criteria:

* Signed informed consent must be obtained prior to the initiation of any study-required procedures. The participant has a parent, caregiver, or legal representative (referred to as "caregiver") who is reliable and able to consent for the participant according to ICH and local regulations

  * At least 18 years of age
  * Willing and able to accompany the participant to clinic visits and be available to the site by phone, email, or other electronic form as needed
  * Is and will likely remain sufficiently knowledgeable of the participant's condition in order to respond to queries as requested.
* Patient had previously signed informed consent for the TANGELO Optional OOE and completed a final safety follow-up visit for the TANGELO Study.
* Participant is able to comply with all requirements including blood draws.
* Participant is able to undergo lumbar puncture (LP) and intrathecal (IT) injection under sedation or anesthesia as deemed appropriate.
* Will comply with requirements regarding contraception and is confirmed by caregiver consent.
* In the opinion and clinical judgement of the Physician, potential benefit outweighs potential risk of continuing rugonersen as an investigational therapy, based on the individual patient's medical history and program eligibility criteria, and judged by the treating physician to still being medically suitable for treatment with rugonersen.

Exclusion Criteria:

* History of clinically significant post lumbar puncture headache of moderate or severe intensity and/or blood patch.
* Hospitalization for any major medical or surgical procedure involving general anesthesia within 12 weeks of screening or planned during treatment.
* Ascertained or presumptive hypersensitivity to the rugonersen or its excipients.
* Permitted sleep medications have not been stable for 4 weeks prior to screening and at time of enrolment.
* Permitted medications for epilepsy have not been stable for 12 weeks prior to screening and at the time of enrolment.
* Prohibited use of antiplatelet or anticoagulant therapy for 2 weeks prior to screening and at the time of enrolment.
* Concurrent psychotropic medications have not been stable for 4 weeks prior to screening and at time of enrolment.
* Concurrent or planned concurrent participation in any clinical trial (including observational, non-drug or non-interventional).
* Previous participation in cellular therapy, gene therapy or gene editing, or any other gene expression modulating clinical trial, such as an antisense oligonucleotide (ASO) treatment other than rugonersen.
* Participation in any other research study with drug or non-drug treatments during this EAP.
* Participants who discontinued participation in the TANGELO Study (BP41674) due to safety reasons are not eligible.

Sex: All
Age Groups: Child, Adult, Older Adult